CLINICAL TRIAL: NCT03613753
Title: A Randomized Phase II Trial of Irinotecan Plus Lobaplatin Versus Irinotecan for the Second-line Treatment of Relapsed Small-cell Lung Cancer
Brief Title: Irinotecan Plus Lobaplatin Versus Irinotecan in the Second-line Treatment of Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ShengFa Su (Other)
Responsible Party: Sponsor-Investigator, ShengFa Su, Professor, Guizhou Medical University
Organization: Guizhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-SCLC-001
Record Dates: First submitted 2018-07-21; First posted 2018-08-03 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Small-cell Lung Cancer
Keywords: relapsed
MeSH Terms: conditions — Small Cell Lung Carcinoma; Recurrence | interventions — Irinotecan; lobaplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Chemotherapy:irinotecan plus lobaplatin
  Interventions: Drug: irinotecan plus lobaplatin
- Arm B (Active Comparator): Chemotherapy:irinotecan
  Interventions: Drug: irinotecan

INTERVENTIONS:
Drug: irinotecan plus lobaplatin — irinotecan plus lobaplatin chemotherapy
  Arms: Arm A
Drug: irinotecan — irinotecan chemotherapy alone
  Arms: Arm B

SUMMARY:
This randomized phase II study compare survival outcomes and toxicity of two chemotherapy regimens (irinotecan plus lobaplatin or irinotecan) for the second-line treatment of recurrent small-cell lung cancer.

DETAILED DESCRIPTION:
The most widely applied first-line treatment mode for small-cell lung cancer (SCLC) patients was chemotherapy as initial treatment. Etoposide with cisplatin or carboplatin were considered the standard first-line regimen in SCLC. As for second-line chemotherapy, single regimen irinotecan or a combined regimen containing irinotecan were one of preferred regiems. While there still is no consensus on second-line therapy. Clinical studies have demonstrated that the combination of irinotecan and carboplatin or cisplatin did not improve outcome in recurrent SCLC patients compared with irinotecan alone. One of the main reasons is that carboplatin or cisplatin has been used in the first-line treatment, and SCLC showed cross-resistance to carboplatin and cisplatin.

Lobaplatin is a platinum complex with DNA alkylating activity that was developed by ASTA Medica (Degussa) for the treatment of cancer. Lobaplatin as the third-generation platinum antineoplastic agent, showed promising antineoplastic effects in variety of preclinical test tumor models, which overcomes some forms of cisplatin or carboplatin resistance in preclinical tumour models. Retrospective studies also have demonstrated the efficacy of Lobaplatin in patients with relapsed SCLC. Thus, we perform this randomized study to compare the efficacy and safety of irinotecan plus lobaplatin versus irinotecan in patients recurrent SCLC.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed SCLC
* Etoposide with cisplatin or carboplatin was first-line chemotherapy in SCLC
* At least 30 days after the completion of first-line chemotherapy
* Either sex, age between 18 to 70 years
* Expected life time ≥ 3 months
* Performance status ECOG grade 0-1. Patients with PS 2 whose general condition is explained by obstructive/bulky disease likely to improve after the first cycle of chemotherapy can be included at the discretion of the local investigator. Patients with PS 2 as a result of comorbid conditions will be excluded.
* Adequate bone marrow and organ function as defined below:

Neutrophils ≥ 1.5 × 109/L, platelets 80 × 109/L, hemoglobin ≥80 g/L; AST and ALT ≤2× the upper limit of the institutional normal range, total bilirubin ≤1.25× the upper limit of the institutional normal range; Creatinineconcentration ≤120 μmol/L

* Had measurable or assessable disease

Exclusion Criteria:

* Concomitant with other malignant disease
* Pregnancy or lactation at the time of enrollment
* Any contraindications for chemotherapy
* Received target therapy or immunotherapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | >4 weeks post treatment
  Tumor Response will be evaluated using the RECIST 1.1 criteria.ORR is Partial response (PR) and complete response (CR).

SECONDARY OUTCOMES:
Treatment toxicities | up to 12 months
  To assess and record nausea, vomiting, hematologic toxicity,and other treantment complications by CTCAE v4.0
Progression-free survival(PFS) | up to 12 months
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Overall survival(OS) | up to 12 months
  Overall survival is defined as the time interval from date of diagnosis to date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: ShengFa Su, PhD,MD, Principal Investigator — The Affiliated Hospital Of Guizhou Medical University
Locations (1):
- The affiliated hospital of Guizhou medical university, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: Undecided